CLINICAL TRIAL: NCT06008977
Title: Exercise to Boost Response to Checkpoint Blockade Immunotherapy
Acronym: EX-BOOST
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: AdventHealth Translational Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 1805426
Record Dates: First submitted 2023-06-06; First posted 2023-08-24 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-06

CONDITIONS: Cutaneous Melanoma; Cutaneous Squamous Cell Carcinoma; Merkel Cell Carcinoma
MeSH Terms: conditions — Melanoma; Carcinoma, Merkel Cell | interventions — Exercise Test

STUDY DESIGN:
Intervention Model Description: We will use stratified block randomization to assure non-biased assignment to the exercise intervention arm. Within each treatment setting, adjuvant and neoadjuvant, 10 patients will be randomized to the exercise intervention arm and 10 to the standard treatment arm. Within the neoadjuvant setting, randomization also will be blocked within disease type.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Standard Group- No Exercise (Adjuvant) (No Intervention): Patients randomized to the standard arm will receive clinical care following AH standards for the patient's disease type and therapeutic setting. This includes history and physical and laboratory studies to be conducted on each infusion day before clearing the patient for infusion.
- Intervention Group- Moderate Exercise (adjuvant) (Active Comparator): Patients randomized to the exercise arm will complete up to 30 minutes of same-day exercise prior to each administration of checkpoint blockade immunotherapy across all cycles. The preferred exercise is 30 minutes of moderate exertion on a cycle ergometer.
  Interventions: Other: Exercise Test
- Standard Group- No Exercise (Neoadjuvant) (No Intervention): Patients randomized to the standard arm will receive clinical care following AH (AdventHealth) standards for the patient's disease type and therapeutic setting. This includes history and physical and laboratory studies to be conducted on each infusion day before clearing the patient for infusion.
- Intervention Group- Moderate Exercise (Neoadjuvant) (Active Comparator): Patients randomized to the exercise arm will complete up to 30 minutes of same-day exercise prior to each administration of checkpoint blockade immunotherapy across all cycles. The preferred exercise is 30 minutes of moderate exertion on a cycle ergometer.
  Interventions: Other: Exercise Test

INTERVENTIONS:
Other: Exercise Test — Supervised pedaling on an ergometer (stationary bike) at a moderate pace for a goal of 30 minutes. The exercise test will be scheduled at infusion visits 1, 6, and 12 or 1 and 3 over the treatment cycle, depending on the group assignment.
  Arms: Intervention Group- Moderate Exercise (Neoadjuvant); Intervention Group- Moderate Exercise (adjuvant)

SUMMARY:
The purpose of this pilot study will be to provide i) information on feasibility implementing an exercise intervention trial among patients with cutaneous cancers, including melanoma, squamous cell carcinoma (cuSCC), and Merkel cell carcinoma, scheduled to receive checkpoint blockade immunotherapy, and ii) preliminary data on the impact of a day-of-therapy exercise intervention.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females ≥18 years of age.
2. Able to read and speak English fluently.
3. Reported ability to complete 20-30 minutes moderate exercise per positive response to, "Can you currently walk unaided for six minutes or more?"
4. Scheduled for first-time checkpoint blockade immunotherapy with avelumab, cemiplimab, ipilimumab, nivolumab, or pembrolizumab in the absence of other therapies (e.g. targeted therapy) with the following diagnosis:

   1. Adjuvant setting: cutaneous melanoma.
   2. Neoadjuvant setting: cutaneous melanoma, cuSCC, or Merkel cell carcinoma.
5. States willingness to follow protocol as described, including the prescribed exercise level and completing any forms needed throughout the study.
6. Voluntarily signed and dated an informed consent form, approved by an Institutional Review Board/Independent Ethics Committee, and provided Health Insurance Portability and Accountability Act authorization (HIPAA) or other privacy authorization prior to any participation in study.

   Exclusion Criteria:
7. Presence of medical conditions, such as severe cardiovascular disease for which exercise may be contraindicated. Participants may be referred to their medical team to obtain a cardiology approval.
8. Presence of major postoperative complications for which an exercise intervention may be contraindicated.
9. Currently has a chronic, contagious, infectious disease, such as active tuberculosis, active Hepatitis B or C, HIV, or COVID-19, per self-report.
10. Currently pregnant, lactating or planning to become pregnant (positive result on urine pregnancy testing).
11. Presence of any condition that, in the opinion of the Investigator, compromises participant safety or data integrity or the participant's ability to complete the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-06-03 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Relapse-free survival | Up to 12 months
  For patients treated in the adjuvant setting. Total study duration is dependent upon oncology therapy.
  Recurrence-free survival will be assessed.
Pathological complete response (pCR) | Up to 12 months
  For patients treated in the neoadjuvant setting. All neoadjuvant patients will have remaining tumor and, when appropriate, its associated nodal basin removed after completion of checkpoint blockade immunotherapy. Total study duration is dependent upon oncology therapy.
  This will be measured in excised tissues after standard-of-care surgery post completion of checkpoint blockade immunotherapy.

CONTACTS AND LOCATIONS:
Overall Officials: Bret Goodpaster, PhD, Principal Investigator — Study Principal Investigator
Locations (1):
- AdventHealth Translational Research Institute, Orlando, Florida, United States

REFERENCES:
- [Background] Hojman P, Gehl J, Christensen JF, Pedersen BK. Molecular Mechanisms Linking Exercise to Cancer Prevention and Treatment. Cell Metab. 2018 Jan 9;27(1):10-21. doi: 10.1016/j.cmet.2017.09.015. Epub 2017 Oct 19. PMID 29056514
- [Background] Campbell JP, Turner JE. Debunking the Myth of Exercise-Induced Immune Suppression: Redefining the Impact of Exercise on Immunological Health Across the Lifespan. Front Immunol. 2018 Apr 16;9:648. doi: 10.3389/fimmu.2018.00648. eCollection 2018. PMID 29713319
- [Background] Martin-Ruiz A, Fiuza-Luces C, Rincon-Castanedo C, Fernandez-Moreno D, Galvez BG, Martinez-Martinez E, Martin-Acosta P, Coronado MJ, Franco-Luzon L, Gonzalez-Murillo A, Ramirez M, Provencio M, Lucia A. Benefits of exercise and immunotherapy in a murine model of human non-small-cell lung carcinoma. Exerc Immunol Rev. 2020;26:100-115. PMID 32139351
- [Background] Montes J, McDermott MP, Martens WB, Dunaway S, Glanzman AM, Riley S, Quigley J, Montgomery MJ, Sproule D, Tawil R, Chung WK, Darras BT, De Vivo DC, Kaufmann P, Finkel RS; Muscle Study Group and the Pediatric Neuromuscular Clinical Research Network. Six-Minute Walk Test demonstrates motor fatigue in spinal muscular atrophy. Neurology. 2010 Mar 9;74(10):833-8. doi: 10.1212/WNL.0b013e3181d3e308. PMID 20211907
- [Background] Tetzlaff MT, Messina JL, Stein JE, Xu X, Amaria RN, Blank CU, van de Wiel BA, Ferguson PM, Rawson RV, Ross MI, Spillane AJ, Gershenwald JE, Saw RPM, van Akkooi ACJ, van Houdt WJ, Mitchell TC, Menzies AM, Long GV, Wargo JA, Davies MA, Prieto VG, Taube JM, Scolyer RA. Pathological assessment of resection specimens after neoadjuvant therapy for metastatic melanoma. Ann Oncol. 2018 Aug 1;29(8):1861-1868. doi: 10.1093/annonc/mdy226. PMID 29945191
- [Background] Weber J, Mandala M, Del Vecchio M, Gogas HJ, Arance AM, Cowey CL, Dalle S, Schenker M, Chiarion-Sileni V, Marquez-Rodas I, Grob JJ, Butler MO, Middleton MR, Maio M, Atkinson V, Queirolo P, Gonzalez R, Kudchadkar RR, Smylie M, Meyer N, Mortier L, Atkins MB, Long GV, Bhatia S, Lebbe C, Rutkowski P, Yokota K, Yamazaki N, Kim TM, de Pril V, Sabater J, Qureshi A, Larkin J, Ascierto PA; CheckMate 238 Collaborators. Adjuvant Nivolumab versus Ipilimumab in Resected Stage III or IV Melanoma. N Engl J Med. 2017 Nov 9;377(19):1824-1835. doi: 10.1056/NEJMoa1709030. Epub 2017 Sep 10. PMID 28891423
- [Background] Khunger A, Buchwald ZS, Lowe M, Khan MK, Delman KA, Tarhini AA. Neoadjuvant therapy of locally/regionally advanced melanoma. Ther Adv Med Oncol. 2019 Jul 31;11:1758835919866959. doi: 10.1177/1758835919866959. eCollection 2019. PMID 31391869
- See also: Website for AdventHealth Translational Research Institute — https://www.adventhealthresearchinstitute.com/research/translational-research